CLINICAL TRIAL: NCT04737863
Title: Minimally Invasive Management of Separated Instruments in Vertucci Type ii Canals: A Radomized Clinical Trial
Brief Title: Minimally Invasive Management During Endodontic Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Mokhtar Nagy, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASFD-ENDO-2
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Teeth, Endodontically-Treated
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selective root canal retreatment (Experimental): retreatment process is performed to the affected root only
  Interventions: Procedure: Endodontic retreatment
- traditional root canal retreatment (Active Comparator): retreatment process is performed to all roots
  Interventions: Procedure: Endodontic retreatment

INTERVENTIONS:
Procedure: Endodontic retreatment — Root canal retreatment in cases with secondary root canal infection

SUMMARY:
The study compares the prognosis of cases treated with "selective root retreatment" to the cases treated with traditional retreatment approach

DETAILED DESCRIPTION:
Post-treatment apical periodontitis is an inflammatory disorder of peri-radicular tissues caused by either persistent or secondary intra-radicular infection .Conventionally, nonsurgical retreatment has been believed to be an ''all or none'' treatment approach in which the endodontist has to remove all restorations from the tooth and to remove the obturation materials from all the canals in order to perform thorough disinfection of the entire root canal system. Nowadays, All operations in the medical field are aimed basically at the conservation of the human body. The alternative concept allows the endodontist to formulate clinical treatment decisions with respect to the presence of periapical pathosis related to individual roots rather than the tooth as a whole.

The literature is lacking the clinical outcome studies dealing with the prognosis of cases treated with "selective root retreatment" concept so the aim of this study was to compare the prognosis of such cases in comparison to the traditional retreatment approach.

ELIGIBILITY:
Inclusion Criteria:

* endodontically treated teeth
* multirooted teeth
* radiographic evidence of periradicular infection related to one root

Exclusion Criteria:

* medically compromised patients
* fused roots
* root resorption
* root fracture

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
volumetric change of periapical lesion size in CBCT | one year
  assessment of healing of periradicular infection in terms of change of the size of periapical lesion in CBCT analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Nagy, PhD, Principal Investigator — Associate professor of Endodontics, Ain Shams University
Locations (1):
- Faculty of Dentistry, Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nudera WJ. Selective Root Retreatment: A Novel Approach. J Endod. 2015 Aug;41(8):1382-8. doi: 10.1016/j.joen.2015.02.035. Epub 2015 Apr 21. PMID 25906919
- [Result] Liang YH, Li G, Wesselink PR, Wu MK. Endodontic outcome predictors identified with periapical radiographs and cone-beam computed tomography scans. J Endod. 2011 Mar;37(3):326-31. doi: 10.1016/j.joen.2010.11.032. PMID 21329816